CLINICAL TRIAL: NCT03098745
Title: Fitting Evaluation of Hydrogel and Silicone Hydrogel Sphere Design Contact Lenses.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CooperVision, Inc. (Industry)
Responsible Party: Sponsor
Organization: CooperVision International Limited (CVIL) (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: EX-MKTG-79
Record Dates: First submitted 2017-03-28; First posted 2017-04-04 (Actual); Results first posted 2019-04-09 (Actual); Last update posted 2019-04-09 (Actual); Status verified 2019-04

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Omafilcon A (Active Comparator): Participants are randomized to wear omafilcon A lens pair bilaterally for 1 hour during the study.
  Interventions: Device: Omafilcon A
- Somofilcon A (Active Comparator): Participants are randomized to wear somofilcon A lens pair bilaterally for 1 hour during the study.
  Interventions: Device: Somofilcon A
- Omafilcon A - Proclear (PC) (Active Comparator): Participants are randomized to wear omafilcon A - PC lens pair bilaterally for 1 hour during the study.
  Interventions: Device: Omafilcon A - Proclear (PC)

INTERVENTIONS:
Device: Omafilcon A — contact lens
  Arms: Omafilcon A
Device: Somofilcon A — contact lens
  Arms: Somofilcon A
Device: Omafilcon A - Proclear (PC) — contact lens
  Arms: Omafilcon A - Proclear (PC)

SUMMARY:
The aim of this non-dispensing fitting study is to evaluate the short term lens fit, vision performance of three monthly replacement sphere lenses.

DETAILED DESCRIPTION:
This is a 40-subject, double masked, randomized, bilateral, non-dispensing fitting trial comparing hydrogel and silicone hydrogel lens materials. It is anticipated that this study will involve 2 visits for each lens pair, as follows: Visits: V1 (lens dispensing), V2 (1 hour post lens settling). Each subject will be randomized to wear each pair bilaterally in a series of three short fitting comparisons.

ELIGIBILITY:
Inclusion Criteria:

* A person is eligible for inclusion in the study if he/she:

  * Is between 18 and 40 years of age (inclusive).
  * Has had a self-reported visual exam in the last two years.
  * Is an adapted soft CL (Contact Lens) wearer who is not wearing any of the study lenses.
  * Has a CL spherical prescription between - 1.00 and - 6.00 (inclusive)
  * Has a spectacle cylinder up to 0.75D (Diopter) in each eye.
  * Can achieve best corrected spectacle distance visual acuity of 20/25 (0.10 logMAR) or better in each eye.
  * Can achieve a distance visual acuity of 20/30 (0.18 logMAR) or better in each eye with the study contact lenses.
  * Has clear corneas and no active ocular disease.
  * Has read, understood and signed the information consent letter.
  * Patient contact lens refraction should fit within the available parameters of the study lenses.
  * Is willing to comply with the wear schedule.
  * Is willing to comply with the visit schedule.

Exclusion Criteria:

* A person will be excluded from the study if he/she:

  * Has never worn contact lenses before.
  * Currently wears rigid gas permeable contact lenses.
  * Has a history of not achieving comfortable CL wear (5 days per week; > 8 hours/day)
  * Has a CL prescription outside the range of - 1.00 to - 6.00D
  * Has a spectacle cylinder ≥1.00D of cylinder in either eye.
  * Has contact lens best corrected distance vision worse than 20/25 (0.10 logMAR) in either eye.
  * Presence of clinically significant (grade 2-4) anterior segment abnormalities.
  * Presence of ocular or systemic disease or need of medications which might interfere with contact lens wear.
  * Slit lamp findings that would contraindicate contact lens wear such as:

    * Pathological dry eye or associated findings
    * Pterygium, pinguecula, or corneal scars within the visual axis
    * Neovascularization > 0.75 mm in from of the limbus
    * Giant papillary conjunctivitis (GCP) worse than grade 1
    * Anterior uveitis or iritis (past or present)
    * Seborrheic eczema, Seborrheic conjunctivitis
    * History of corneal ulcers or fungal infections
    * Poor personal hygiene
  * Has a known history of corneal hypoesthesia (reduced corneal sensitivity)
  * Has aphakia, keratoconus or a highly irregular cornea.
  * Has Presbyopia or has dependence on spectacles for near work over the contact lenses.
  * Has undergone corneal refractive surgery.
  * Is participating in any other type of eye related clinical or research study.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2017-03-01 (Actual); Study Completion 2017-04-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ruben Velázquez Guerrero, MSc., FIACLE, Principal Investigator — National Autonomous University, School of Optometry
Locations (1):
- Optometry Clinic, National Autonomous University, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Omafilcon A, Omafilcon A - Proclear (PC), Somofilcon A: Participants are randomized to wear omafilcon A lens pair bilaterally for 1 hour during this double masked nondispensing fitting study, then omafilcon A - Proclear (PC), then Somofilcon A lens pair bilaterally for 1 hour.
- Omafilcon A, Somofilcon A, Omafilcon A - Proclear (PC): Participants are randomized to wear omafilcon A lens pair bilaterally for 1 hour during this double masked nondispensing fitting study, then Somofilcon A, then omafilcon A - Proclear (PC) lens pair bilaterally for 1 hour.
- Somofilcon A, Omafilcon A - Proclear (PC), Omafilcon A: Participants are randomized to wear somofilcon A lens pair bilaterally for 1 hour during this double masked nondispensing fitting study, then omafilcon A - Proclear (PC), then omafilcon A lens pair bilaterally for 1 hour.
- Somofilcon A, Omafilcon A, Omafilcon A- Proclear (PC): Participants are randomized to wear somofilcon A lens pair bilaterally for 1 hour during this double masked nondispensing fitting study, then omafilcon A, then omafilcon A - Proclear (PC) lens pair bilaterally for 1 hour.
- Omafilcon A - Proclear (PC), Omafilcon A, Somofilcon A: Participants are randomized to wear omafilcon A - Proclear (PC) lens pair bilaterally for 1 hour during this double masked nondispensing fitting study, then omafilcon A, then somofilcon A lens pair bilaterally for 1 hour.
- Omafilcon A - Proclear (PC), Somofilcon A, Omafilcon A: Participants are randomized to wear omafilcon A - Proclear (PC) lens pair bilaterally for 1 hour during this double masked nondispensing fitting study, then somofilcon A, then omafilcon A lens pair bilaterally for 1 hour.
Period: Day 1
Arm/Group | Omafilcon A, Omafilcon A - Proclear (PC), Somofilcon A | Omafilcon A, Somofilcon A, Omafilcon A - Proclear (PC) | Somofilcon A, Omafilcon A - Proclear (PC), Omafilcon A | Somofilcon A, Omafilcon A, Omafilcon A- Proclear (PC) | Omafilcon A - Proclear (PC), Omafilcon A, Somofilcon A | Omafilcon A - Proclear (PC), Somofilcon A, Omafilcon A
Started | 7 | 3 | 8 | 8 | 10 | 4
Completed | 7 | 3 | 8 | 8 | 10 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Day 2
Arm/Group | Omafilcon A, Omafilcon A - Proclear (PC), Somofilcon A | Omafilcon A, Somofilcon A, Omafilcon A - Proclear (PC) | Somofilcon A, Omafilcon A - Proclear (PC), Omafilcon A | Somofilcon A, Omafilcon A, Omafilcon A- Proclear (PC) | Omafilcon A - Proclear (PC), Omafilcon A, Somofilcon A | Omafilcon A - Proclear (PC), Somofilcon A, Omafilcon A
Started | 7 | 3 | 8 | 8 | 10 | 4
Completed | 7 | 3 | 8 | 8 | 10 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Day 3
Arm/Group | Omafilcon A, Omafilcon A - Proclear (PC), Somofilcon A | Omafilcon A, Somofilcon A, Omafilcon A - Proclear (PC) | Somofilcon A, Omafilcon A - Proclear (PC), Omafilcon A | Somofilcon A, Omafilcon A, Omafilcon A- Proclear (PC) | Omafilcon A - Proclear (PC), Omafilcon A, Somofilcon A | Omafilcon A - Proclear (PC), Somofilcon A, Omafilcon A
Started | 7 | 3 | 8 | 8 | 10 | 4
Completed | 7 | 3 | 8 | 8 | 10 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Overall Study: Participants are randomized to wear omafilcon A lens pair, Somofilcon A lens pair, Omafilcon A - Proclear PC bilaterally for 1 hour during the study on separate days
Arm/Group | Overall Study
Number analyzed (Participants) | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 40
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.3 (6.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30
  Male | 10
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Mexico | 40

OUTCOME MEASURES:

1. Primary Outcome: Visual Acuity
Description: High contrast distance visual acuity assessed for each lens pair using LogMAR chart at time of lens insertion, then assessing again 1 hour later with spectacles after lenses are removed.
Time Frame: Baseline (lens insertion), 1 hour
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | Omafilcon A | Somofilcon A | Omafilcon A - Proclear (PC)
Number analyzed (Participants) | 40 | 40 | 40
logMAR
  Lens Insertion (CL) | -0.04 (0.05) | -0.05 (0.05) | -0.03 (0.04)
  1 Hour (Specs) | -0.01 (0.03) | -0.01 (0.03) | -0.01 (0.02)

2. Primary Outcome: Comfort
Description: Subjective comfort (Scale 0-100: 0=very uncomfortable, 100= very comfortable)
Time Frame: Insertion, 1hr
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Omafilcon A | Somofilcon A | Omafilcon A - Proclear (PC)
Number analyzed (Participants) | 40 | 40 | 40
units on a scale
  Insertion | 94.5 (8.5) | 98.0 (5.0) | 94.7 (7.4)
  1 Hour | 95.8 (8.2) | 96.8 (5.5) | 93.7 (10.7)

3. Primary Outcome: Lens Centration
Description: Centration of lens on eye (Scale: Optimum, Decentration acceptable, Decentration unacceptable)
Time Frame: Insertion
Measure: Count of Participants; unit: Participants
Arm/Group | Omafilcon A | Somofilcon A | Omafilcon A - Proclear (PC)
Number analyzed (Participants) | 40 | 40 | 40
Participants
  Optimum | 40 | 40 | 40
  Decentration Acceptable | 0 | 0 | 0
  Decentration Unacceptable | 0 | 0 | 0

4. Primary Outcome: Lens Centration
Description: Centration of lens on eye (Scale: Optimum, Decentration acceptable, Decentration unacceptable)
Time Frame: 1 Hour
Measure: Count of Participants; unit: Participants
Arm/Group | Omafilcon A | Somofilcon A | Omafilcon A - Proclear (PC)
Number analyzed (Participants) | 40 | 40 | 40
Participants
  Optimum | 40 | 40 | 40
  Decentration Acceptable | 0 | 0 | 0
  Decentration Unacceptable | 0 | 0 | 0

5. Primary Outcome: Post-blink Lens Movement
Description: Amount of lens movement after blink (Scale: Insufficient, Minimum, Optimum, Moderate, Excessive)
Time Frame: Insertion
Measure: Count of Participants; unit: Participants
Arm/Group | Omafilcon A | Somofilcon A | Omafilcon A - Proclear (PC)
Number analyzed (Participants) | 40 | 40 | 40
Participants
  Insufficient | 1 | 0 | 1
  Minimum | 9 | 1 | 7
  Optimum | 27 | 31 | 19
  Moderate | 3 | 8 | 13
  Excessive | 0 | 0 | 0

6. Primary Outcome: Post-blink Lens Movement
Description: Amount of lens movement after blink (Scale: Insufficient, Minimum, Optimum, Moderate, Excessive)
Time Frame: 1 Hour
Measure: Count of Participants; unit: Participants
Arm/Group | Omafilcon A | Somofilcon A | Omafilcon A - Proclear (PC)
Number analyzed (Participants) | 40 | 40 | 40
Participants
  Insufficient | 0 | 1 | 0
  Minimum | 7 | 1 | 4
  Optimum | 31 | 37 | 34
  Moderate | 2 | 1 | 2
  Excessive | 0 | 0 | 0

7. Primary Outcome: Lens Fit Acceptance
Description: Investigator's determination of whether lens fit is acceptable (Scale: Shouldn't be worn, Borderline, Min Acceptable, OK to dispense, Perfect)
Time Frame: Insertion
Measure: Count of Participants; unit: Participants
Arm/Group | Omafilcon A | Somofilcon A | Omafilcon A - Proclear (PC)
Number analyzed (Participants) | 40 | 40 | 40
Participants
  Shouldn't be worn | 0 | 0 | 1
  Borderline | 2 | 2 | 4
  Min acceptable | 2 | 1 | 3
  OK to dispense | 10 | 8 | 10
  Perfect | 26 | 29 | 22

8. Primary Outcome: Lens Fit Acceptance
Description: as for outcome 7
Time Frame: 1 Hour
Measure: Count of Participants; unit: Participants
Arm/Group | Omafilcon A | Somofilcon A | Omafilcon A - Proclear (PC)
Number analyzed (Participants) | 40 | 40 | 40
Participants
  Shouldn't be worn | 0 | 1 | 0
  Borderline | 0 | 0 | 4
  Min acceptable | 5 | 1 | 0
  OK to dispense | 5 | 3 | 3
  Perfect | 30 | 35 | 33

9. Primary Outcome: Lens Fit Preference
Description: Investigator lens fit preference (Scale: omafilcon A, somofilcon A, omafilcon A - Proclear (PC))
Time Frame: 1 Hour
Measure: Count of Participants; unit: Participants
Groups:
- Overall Study: Investigator's preference of lens based on fit
Arm/Group | Overall Study
Number analyzed (Participants) | 40
Participants
  omafilcon A | 5
  somofilcon A | 2
  omafilcon A - Proclear (PC) | 6
  No Preference | 27

10. Primary Outcome: Limbal Redness
Description: Redness of limbal area (Scale: 0-4, 0 = none, 4=severe)
Time Frame: 1 Hour
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Omafilcon A | Somofilcon A | Omafilcon A - Proclear (PC)
Number analyzed (Participants) | 40 | 40 | 40
units on a scale | 0.41 (0.3) | 0.39 (0.3) | 0.39 (0.3)

11. Primary Outcome: Bulbar Redness
Description: Redness of bulbar conjunctiva (Scale: 0-4, 0 = none, 4=severe)
Time Frame: 1 Hour
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Omafilcon A | Somofilcon A | Omafilcon A - Proclear (PC)
Number analyzed (Participants) | 40 | 40 | 40
units on a scale | 0.51 (0.36) | 0.55 (0.38) | 0.50 (0.37)

ADVERSE EVENTS:
Time Frame: 1 hour visit
Arm/Group | Omafilcon A | Somofilcon A | Omafilcon A - Proclear (PC)
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/40 | 0/40
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/40 | 0/40
Other Adverse Events (participants affected / at risk) | 0/40 | 0/40 | 0/40

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-01-13): https://cdn.clinicaltrials.gov/large-docs/45/NCT03098745/Prot_SAP_000.pdf